CLINICAL TRIAL: NCT03402386
Title: A Phase III, Open-label Study of MT-6548 in Peritoneal Dialysis Subjects With Anemia Associated With Chronic Kidney Disease in Japan
Brief Title: Efficacy and Safety Study to Evaluate MT-6548 in Peritoneal Dialysis Subjects With Anemia Associated With Chronic Kidney Disease in Japan
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Tanabe Pharma Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MT-6548-J02
Record Dates: First submitted 2017-12-27; First posted 2018-01-18 (Actual); Results first posted 2021-07-06 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2025-12

CONDITIONS: Anemia; Peritoneal Dialysis Dependent Chronic Kidney Disease
MeSH Terms: conditions — Anemia | interventions — vadadustat

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- MT-6548 (Experimental)
  Interventions: Drug: MT-6548

INTERVENTIONS:
Drug: MT-6548 — Oral tablet
  Other Names: vadadustat; AKB-6548

SUMMARY:
To evaluate the efficacy and safety of MT-6548 in peritoneal dialysis subjects with anemia associated with chronic kidney disease

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of CKD
* Receiving peritoneal dialysis for more than 4 weeks prior to the screening period. However, receiving hemodialysis is excluded
* Not expected to start hemodialysis during the study
* Correction group: Not being treated with ESAs for the recent 8 weeks prior to the screening period
* Conversion group: Being treated with ESAs for the recent 8 weeks prior to the screening period
* Mean of the two screening Hb levels closest in time to the baseline visit. Correction group: ≥8.0 g/dL and < 11.0 g/dL Conversion group: ≥9.0 g/dL and ≤12.5 g/dL
* Fluctuation between the two Hb levels closest in time to the baseline visit during the screening period less than 1.5 g/dL
* Serum ferritin ≥ 100 ng/mL, or TSAT ≥20% during the screening period
* Folate and vitamin B12 ≥ lower limit of normal during the screening period

Exclusion Criteria:

* Anemia due to a main cause other than CKD: sickle cell disease, myelodysplastic syndrome, bone marrow fibrosis, hematologic malignancy, hemolytic anemia, thalassemia, or pure red cell aplasia
* Active bleeding or recent blood loss within 8 weeks prior to the screening period
* RBC transfusion within 8 weeks prior to the screening period
* Received testosterone enanthate or mepitiostane within 8 weeks prior to the screening period
* Peritonitis within 4 weeks prior to the screening period
* AST, ALT, or total bilirubin >2.5 x upper limit of normal during the screening period
* Uncontrolled hypertension (diastolic blood pressure >110 mm Hg or systolic blood pressure >180 mm Hg) during the screening period and Day 1
* Ophthalmic examinations during the screening period correspond to either of the following criteria;

  * No available fundal findings
  * Findings indicating the presence of active fundal disease
* Severe heart failure (New York Heart Association Class IV)
* Cerebrovascular disorder or acute coronary syndrome (e.g. hospitalization due to unstable angina or myocardial infarction), requiring hospitalization due to urgent percutaneous intervention for coronary or heart failure within 12 weeks prior to the screening period
* Current or history of malignancy. History of malignancy with no recurrence for the recent 5 years is not an exclusion criterion
* New onset or recurrent event of deep vein thrombosis or pulmonary embolism within 12 weeks prior to the screening period
* Current or history of hemosiderosis or hemochromatosis
* History of prior organ transplantation or scheduled organ transplant, or prior transplantation of hematopoietic stem cell or bone marrow
* Males and females of childbearing potential who are unwilling to use an acceptable method of contraception during the designated period (Males: during the study and 90 days after the last dose, Females: during study and 30 days after the last dose)
* Females who are pregnant or breast feeding, or are predicted to be pregnant

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2018-01-03 (Actual); Primary Completion 2018-11-22 (Actual); Study Completion 2018-12-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: General Manager, Study Director — Tanabe Pharma Corporation
Locations (17):
- Japan (17):
  - Research site, Aichi
  - Research site, Chiba
  - Research site, Fukuoka
  - Research site, Fukushima
  - Research site, Gunma
  - Research site, Hokkaido
  - Research site, Hyōgo
  - Research site, Ibaraki
  - Research site, Kagoshima
  - Research site, Kanagawa
  - Research site, Kyoto
  - Research site, Nagano
  - Research site, Nara
  - Research site, Okayama
  - Research site, Okinawa
  - Research site, Shiga
  - Research site, Tokyo

REFERENCES:
- [Result] Nangaku M, Kondo K, Takabe S, Ueta K, Kaneko G, Otsuka M, Kawaguchi Y, Komatsu Y. Vadadustat for anemia in chronic kidney disease patients on peritoneal dialysis: A phase 3 open-label study in Japan. Ther Apher Dial. 2021 Oct;25(5):642-653. doi: 10.1111/1744-9987.13611. Epub 2020 Dec 29. PMID 33283981

RESULTS

PARTICIPANT FLOW:
Groups:
- MT-6548: MT-6548: Oral tablet. The dose was adjusted to 150-600 mg/day according to the pre-specified dose adjustment algorithm.
Period: Overall Study
Arm/Group | MT-6548
Started | 42
Correction Group | 2
Conversion Group | 40
Completed | 36
Not Completed | 6
Not completed — Adverse Event | 3
Not completed — Physician Decision | 1
Not completed — Difficult to control Hb | 2

BASELINE CHARACTERISTICS:
Arm/Group | MT-6548
Number analyzed (Participants) | 42
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 19
  >=65 years | 23
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12
  Male | 30
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian (Japanese) | 42
  Asian (Other) | 0
  Other | 0

OUTCOME MEASURES:

1. Primary Outcome: Mean Hb Level of Week 20 and Week 24
Time Frame: Up to Week 24
Population: This analysis was performed in subjects who measured Hb at least one visit after baseline.
Measure: Least Squares Mean (95% Confidence Interval); unit: g/dL
Arm/Group | MT-6548
Number analyzed (Participants) | 41
g/dL | 11.35 [10.99 to 11.70]

2. Primary Outcome: Hb Level at Each Assessment Time Point
Time Frame: Up to Week 24
Population: This analysis was performed only in subjects who have Hb data at each visit.
Measure: Mean (95% Confidence Interval); unit: g/dL
Arm/Group | MT-6548
Number analyzed (Participants) | 42
g/dL
  Baseline | 10.90 [10.56 to 11.25]
  Week 2: number analyzed (Participants) | 40
  Week 2 | 10.96 [10.54 to 11.38]
  Week 4: number analyzed (Participants) | 41
  Week 4 | 10.74 [10.31 to 11.17]
  Week 6: number analyzed (Participants) | 39
  Week 6 | 10.61 [10.09 to 11.13]
  Week 8: number analyzed (Participants) | 38
  Week 8 | 10.87 [10.41 to 11.33]
  Week 10: number analyzed (Participants) | 38
  Week 10 | 10.89 [10.45 to 11.32]
  Week 12: number analyzed (Participants) | 38
  Week 12 | 11.10 [10.67 to 11.53]
  Week 16: number analyzed (Participants) | 37
  Week 16 | 11.58 [11.12 to 12.04]
  Week 20: number analyzed (Participants) | 36
  Week 20 | 11.68 [11.24 to 12.13]
  Week 24: number analyzed (Participants) | 35
  Week 24 | 11.39 [11.00 to 11.79]
  Week 24 (LOCF): number analyzed (Participants) | 41
  Week 24 (LOCF) | 11.01 [10.54 to 11.47]

3. Primary Outcome: Percentage of Subjects With Hb Level at Each Assessment Time Point Within the Target Range During the Treatment Period
Time Frame: Up to Week 24
Population: This analysis was performed only in subjects who have Hb data at each visit.
Measure: Number; unit: percentage of subjects
Arm/Group | MT-6548
Number analyzed (Participants) | 42
percentage of subjects
  Baseline | 57.1
  Week 2: number analyzed (Participants) | 40
  Week 2 | 60.0
  Week 4: number analyzed (Participants) | 41
  Week 4 | 41.5
  Week 6: number analyzed (Participants) | 39
  Week 6 | 35.9
  Week 8: number analyzed (Participants) | 38
  Week 8 | 47.4
  Week 10: number analyzed (Participants) | 38
  Week 10 | 44.7
  Week 12: number analyzed (Participants) | 38
  Week 12 | 44.7
  Week 16: number analyzed (Participants) | 37
  Week 16 | 32.4
  Week 20: number analyzed (Participants) | 36
  Week 20 | 66.7
  Week 24: number analyzed (Participants) | 35
  Week 24 | 65.7

4. Primary Outcome: Time to Reach the Target Hb Range in Correction Group Only
Time Frame: Up to Week 24
Population: The target number of subjects by correction and conversion group was not pre-specified in the study protocol, and only 2 subjects were enrolled in the correction group as a result. The reason no data have been shown in this column is that this planned analysis wasn't performed due to such insufficient and very small amount of data from the correction group.
Arm/Group | MT-6548
Number analyzed (Participants) | 0

5. Primary Outcome: Rate of Increase in Hb Level in Correction Group Only
Time Frame: Up to Week 6
Population: as for outcome 4
Arm/Group | MT-6548
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: 24 weeks
Arm/Group | MT-6548
All-Cause Mortality (participants affected / at risk) | 1/42
Serious Adverse Events (participants affected / at risk) | 12/42
Other Adverse Events (participants affected / at risk) | 21/42
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | MT-6548 (N=42)
Anaemia (Blood and lymphatic system disorders) | 1
Cardiac failure chronic (Cardiac disorders) | 1
Myocardial ischaemia (Cardiac disorders) | 1
Gastric polyps (Gastrointestinal disorders) | 1
Inguinal hernia (Gastrointestinal disorders) | 1
Catheter site infection (Infections and infestations) | 1
Peritonitis (Infections and infestations) | 3
Sepsis (Infections and infestations) | 1
Peritoneal dialysis complication (Injury, poisoning and procedural complications) | 1
Shunt occlusion (Injury, poisoning and procedural complications) | 1
Traumatic haemothorax (Injury, poisoning and procedural complications) | 1
Cerebral infarction (Nervous system disorders) | 1
Peripheral arterial occlusive disease (Vascular disorders) | 2
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | MT-6548 (N=42)
Abdominal pain upper (Gastrointestinal disorders) | 3
Diarrhoea (Gastrointestinal disorders) | 8
Nausea (Gastrointestinal disorders) | 3
Vomiting (Gastrointestinal disorders) | 4
Catheter site infection (Infections and infestations) | 9
Nasopharyngitis (Infections and infestations) | 6
Decreased appetite (Metabolism and nutrition disorders) | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (2):
  • Study Protocol (2017-12-26): https://cdn.clinicaltrials.gov/large-docs/86/NCT03402386/Prot_000.pdf
  • Statistical Analysis Plan (2019-03-26): https://cdn.clinicaltrials.gov/large-docs/86/NCT03402386/SAP_001.pdf